CLINICAL TRIAL: NCT03865485
Title: RISE- Prevention of Child Mental Health Problems in Southeastern Europe - Adapt, Optimize, Test and Extend Parenting for Lifelong Health - A Factorial Study (Phase 2 of MOST)
Brief Title: Prevention of Child Mental Health Problems in Southeastern Europe (RISE) - A Factorial Study (Phase 2 of MOST)
Acronym: RISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bremen (Other)
Collaborators: University of Klagenfurt (Other); University of Oxford (Other); Bangor University (Other); Babes-Bolyai University (Other); Institute for Marriage, Family and Systemic Practice - ALTERNATIVA (Other); Health for Youth Association, Moldova (Other); University of Cape Town (Other); Georgia State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: H2020-779318; H2020-SC1-2017-RTD-779318 (Other Grant/Funding Number: European Commission)
Record Dates: First submitted 2019-02-25; First posted 2019-03-07 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-04

CONDITIONS: Child Mental Disorder
Keywords: Parenting Program
MeSH Terms: conditions — Neurodevelopmental Disorders

STUDY DESIGN:
Intervention Model Description: Factorial Assignment For the study, a factorial design will be used testing 3 components. With these three components, there will be a total of eight conditions. The purpose of this factorial experiment is to estimate the main effects of the three intervention components and interactions between the components, not to compare the 8 experimental conditions to each other. Each main effect and interaction estimate is based on all of the experimental conditions.
Who Masked: Participant, Investigator
Masking Description: The implementing partners in each country site will notify the participating families of their allocation status (based on clusters) after baseline data collection is completed in each cluster to assure that participants are blind to allocation during the initial assessment. Research assistants conducting data assessments and conducting analysis will be blind to allocation to minimize assessment bias. Because of facilitators' involvement in the program implementation, blinding will not be possible for service providers. Similarly, participants will not be blind to their own treatment condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Length: long; Engagement booster: high; Fidelity booster: high (Experimental): Behavioral: Parenting for Lifelong Health (PLH)
  1. Program length - long: 10 group sessions of the PLH 2-9 intervention delivered every other week (i.e., relationship building, positive reinforcement, setting limits, and effective discipline);
  2. Engagement booster - high: Engagement Boosters (i.e., a communication booster including weekly text messages reminders and 5-minute phone consultations twice a month from facilitators and an enhanced incentives package (including lunch (approx. 1-3€), a food parcel (approx. 2 - 5 €), reimbursement for local transport (FYR of Macedonia and Republic of Moldova only) at each group session and an award for attendance (if parents did not miss more than 1 session, approx. 5-20€) and raffle prizes at the end of the program),
  3. Fidelity booster - high supervision: Fidelity Boosters (i.e., 5 structured intensive video feedback supervision sessions for facilitators).
  Interventions: Behavioral: Parenting for Lifelong Health (PLH)
- Length: long; Engagement booster: high; Fidelity booster: low (Experimental): Behavioral: Parenting for Lifelong Health (PLH)
  1. Program length - long: 10 group sessions of the PLH 2-9 intervention delivered every other week (i.e., relationship building, positive reinforcement, setting limits, and effective discipline);
  2. Engagement booster - high: Engagement Boosters (i.e., a communication booster including weekly text messages reminders and 5-minute phone consultations twice a month from facilitators and an enhanced incentives package (including lunch (approx. 1-3€), a food parcel (approx. 2 - 5 €), reimbursement for local transport (FYR of Macedonia and Republic of Moldova only) at each group session and an award for attendance (if parents did not miss more than 1 session, approx. 5-20€) and raffle prizes at the end of the program),
  3. Fidelity booster - low supervision: No Fidelity Boosters (i.e., supervision on demand only).
  Interventions: Behavioral: Parenting for Lifelong Health (PLH)
- Length: long; Engagement booster: low; Fidelity booster: high (Experimental): Behavioral: Parenting for Lifelong Health (PLH)
  1. Program length - long: 10 group sessions of the PLH 2-9 intervention delivered every other week (i.e., relationship building, positive reinforcement, setting limits, and effective discipline);
  2. Engagement booster - low: No Engagement Boosters
  3. Fidelity booster - high supervision: Fidelity Boosters (i.e., 5 structured intensive video feedback supervision sessions for facilitators).
  Interventions: Behavioral: Parenting for Lifelong Health (PLH)
- Length: long; Engagement booster: low; Fidelity booster: low (Experimental): Behavioral: Parenting for Lifelong Health (PLH)
  1. Program length - long: 10 group sessions of the PLH 2-9 intervention delivered every other week (i.e., relationship building, positive reinforcement, setting limits, and effective discipline);
  2. Engagement booster - low: No Engagement Boosters;
  3. Fidelity booster - low supervision: No Fidelity Boosters (i.e., supervision on demand only).
  Interventions: Behavioral: Parenting for Lifelong Health (PLH)
- Length: short; Engagement booster: high; Fidelity booster:high (Experimental): Behavioral: Parenting for Lifelong Health (PLH)
  1. Program length - short: 5 group sessions of the PLH 2-9 intervention delivered every other week (i.e., relationship building, positive reinforcement, setting limits, and effective discipline);
  2. Engagement booster - high: Engagement Boosters (i.e., a communication booster including weekly text messages reminders and 5-minute phone consultations twice a month from facilitators and an enhanced incentives package (including lunch (approx. 1-3€), a food parcel (approx. 2 - 5 €), reimbursement for local transport (FYR of Macedonia and Republic of Moldova only) at each group session and an award for attendance (if parents did not miss more than 1 session, approx. 5-20€) and raffle prizes at the end of the program),
  3. Fidelity booster - high supervision: Fidelity Boosters (i.e., 5 structured intensive video feedback supervision sessions for facilitators).
  Interventions: Behavioral: Parenting for Lifelong Health (PLH)
- Length: short; Engagement booster: high; Fidelity booster: low (Experimental): Behavioral: Parenting for Lifelong Health (PLH)
  1. Program length - short: 5 group sessions of the PLH 2-9 intervention delivered every other week (i.e., relationship building, positive reinforcement, setting limits, and effective discipline);
  2. Engagement booster - high: Engagement Boosters (i.e., a communication booster including weekly text messages reminders and 5-minute phone consultations twice a month from facilitators and an enhanced incentives package (including lunch (approx. 1-3€), a food parcel (approx. 2 - 5 €), reimbursement for local transport (FYR of Macedonia and Republic of Moldova only) at each group session and an award for attendance (if parents did not miss more than 1 session, approx. 5-20€) and raffle prizes at the end of the program),
  3. Fidelity booster - low supervision: No Fidelity Boosters (i.e., supervision on demand only).
  Interventions: Behavioral: Parenting for Lifelong Health (PLH)
- Length: short; Engagement booster: low; Fidelity booster: high (Experimental): Behavioral: Parenting for Lifelong Health (PLH)
  1. Program length - short: 5 group sessions of the PLH 2-9 intervention delivered every other week (i.e., relationship building, positive reinforcement, setting limits, and effective discipline);
  2. Engagement booster - low: No Engagement Boosters
  3. Fidelity booster - high supervision: Fidelity Boosters (i.e., 5 structured intensive video feedback supervision sessions for facilitators).
  Interventions: Behavioral: Parenting for Lifelong Health (PLH)
- Length: short; Engagement booster: low; Fidelity booster: low (Experimental): Behavioral: Parenting for Lifelong Health (PLH)
  1. Program length - short: 5 group sessions of the PLH 2-9 intervention delivered every other week (i.e., relationship building, positive reinforcement, setting limits, and effective discipline);
  2. Engagement booster - low: No Engagement Boosters
  3. Fidelity booster - low supervision: No Fidelity Boosters (i.e., supervision on demand only).
  Interventions: Behavioral: Parenting for Lifelong Health (PLH)

INTERVENTIONS:
Behavioral: Parenting for Lifelong Health (PLH) — The Parenting for Lifelong Health (PLH) initiative is focused on the development, evaluation, and dissemination of parenting programs to reduce violence against children and improve child wellbeing in LMIC. It was established to address the need to develop low-cost, evidence-based parenting programs that can be integrated within existing service delivery systems in LMIC. The PLH for Young Children from 2-9 y. (PLH 2-9) program includes general content like one-on-one time/child-led play; praising and rewarding children; instructions, household rules, and routines; managing difficult behaviours: ignore and consequences; reflection and moving on. Core activities during sessions include group discussions illustrated vignettes, role-plays, collaborative problem solving, practicing skills at home.

SUMMARY:
The aim of this study is to optimize an adapted version of a parenting program, Parenting for Lifelong Health for Young Children (PLH), to meet the specific needs of families in three low- and middle-income countries in Southeastern Europe (Romania, FYR of Macedonia and Republic of Moldova) using a cluster factorial experimental design to select the most efficacious, cost-effective, and scalable intervention components. This study is the second phase of a three-phase research project (www.rise-plh.eu).

The cluster factorial experiment will examine the effectiveness, cost-effectiveness, and implementation of three selected components of the PLH for Children program to inform the selection of the most effective, cost-effective, and implementable components to include in a prevention package prior to testing it in a subsequent RCT. The cluster factorial experiment will be conducted across three Southeastern European country sites. Each site will recruit families with children aged two to nine years who have elevated levels of child behavior problems, including specifically high-risk groups, such as minorities (e.g. Roma families). Program facilitators will be recruited from local agencies and schools. The factorial experimental trial will randomize 16 clusters in each country to one of 8 experimental conditions which consist of any combination of the three components (program length: 5 sessions/10 sessions; engagement booster: high/low; fidelity booster: high supervision/low supervision). The purpose of this factorial experiment is to estimate the main effects of the three intervention components and interactions between the components.

At the end of the cluster factorial experiment, we will develop an optimized version of the program by selecting components or component levels that have the highest level of effectiveness as based on effect size (rather than p-values). We will also take into consideration factors regarding cost-effectiveness and implementation outcomes when designing this optimized intervention package.

DETAILED DESCRIPTION:
Over the past decade there have been increasing calls for the scale-up of evidence-based interventions in order to reduce the risk of violence against children in low- and middle-income countries (LMICs). In particular, group-based parenting programs for families with young children have been shown to be effective in reducing the risk of child maltreatment and improving child wellbeing with promising evidence emerging from low- and middle-income countries. These group-based programs typically aim to strengthen caregiver-child relationships through positive parenting and help parents to manage child behavior problems through effective, age-appropriate, nonviolent discipline strategies.

Despite the emerging evidence of the effectiveness of parenting interventions in reducing violence against children, many local governments and service providers in LMICs face multiple challenges in implementing evidence-based parenting programs in resource poor contexts. Parenting programs are often too expensive to deliver effectively at scale in low-resource settings due to their complexity, intensity, and length. Parenting programs developed and evaluated in other contexts also may not fit the local service delivery context and may require adaptation to be relevant to the local culture of families. Additional program content may also be necessary to address acute economic deprivation, high community violence, and parental distress. The process of delivery may also need to be simplified to improve participant engagement and the quality of delivery.

As a result, it is essential that programs implemented in LMICs are

1. Effective at reducing violence against children,
2. Integrated within the existing service delivery system of the country,
3. Feasible and culturally acceptable to service providers and families, and
4. Scalable in terms of their affordability, replicability, and sustainability while reaching a maximum number of beneficiaries.

However, there are currently very few parenting programs that meet these criteria in LMICs (such as Romania, FYR of Macedonia and Republic of Moldova), where the need is the greatest.

The Parenting for Lifelong Health (PLH) initiative is focused on the development, evaluation, and dissemination of parenting programs to reduce violence against children and improve child wellbeing in LMIC. It was established to address the need to develop low-cost, evidence-based parenting programs that can be integrated within existing service delivery systems in LMIC. The PLH for Young Children from 2-9 y. (PLH 2-9) program includes general content like one-on-one time/child-led play; praising and rewarding children; instructions, household rules, and routines; managing difficult behaviours: ignore and consequences; reflection and moving on. Core activities during sessions include group discussions illustrated vignettes, role-plays, collaborative problem solving, practicing skills at home.

The present study utilizes the Multiphase Optimization Strategy (MOST) and RE-AIM framework for increasing the reach and enhancing the implementation of PLH 2-9 in three Southeastern European countries with restricted resources. The MOST framework is implemented over 3 distinct phases: 1) Preparation, 2) Optimization, and 3) Evaluation.

The overall RISE project has two general objectives: (1) the first objective relates to the adaption, optimizing and evaluation of selected best practice intervention condition (MOST), while (2) the second objective relates to implementation issues (RE-AIM).

This presently registered study relates to the Optimization Phase (phase 2). This cluster factorial experiment is to inform the selection of the most effective and cost-effective components to include in a prevention package prior to testing in the subsequent RCT.

The factorial experiment will be conducted across the three countries in Southeastern European country sites (N = 48 clusters, 288 families per country site). The study will focus on the recruitment of families from LMICs with children aged two to nine years who have elevated child behaviour problems as well as high-risk groups, i.e. such as Roma families. Program facilitators (N = 80; 16 in FYR of Macedonia, 32 in Republic of Moldova, and in 32 Romania) will be recruited from local agencies and schools. Program coaches (N = 11; 3 in FYR of Macedonia, 4 in Republic of Moldova, and in 4 Romania) will be selected from personnel who previously implemented the PLH 2-9 program during Phase 1.

The following intervention components have been selected (the three components are related to program implementation and efficacy):

Component 1: Engagement booster (high/low): Half of the participants will receive a communication booster (including weekly text messages reminders and 5-minute phone consultations twice a month from facilitators) and an enhanced incentives package (including lunch @ approx. 2-4 euros/person, transport to group sessions when necessary (FYR of Macedonia, and Republic of Moldova only), raffle prize @ approx. 5 euros/person, food parcels @ approx. 2-5 euros/person, and reward for attending all or all but one sessions @ approx. 3-5 euros/person) and half will not receive any engagement boosters. All participants, regardless of condition, will receive a basic incentive package (including child care and a snack) at each group session.

Component 2: Program Length (long: 10 sessions; short: 5 sessions): Half of the participants will receive 5 group sessions (i.e., 10 hours of program delivery and half of the participants will receive 10 group sessions (i.e., 20 hours of program delivery). Both short and long versions will contain the same content as each other and be delivered over the same time period (weekly for the 10 session and fortnightly for the 5 session).

Component 3: Fidelity booster (high supervision/low supervision): Half of the facilitators will receive facilitator training workshop (3-5 days) plus a structured weekly supervision session by a local coach including video feedback (high supervision), while half of the facilitators receive the facilitator training workshop and supervision only upon request (low supervision; low component level).

With this number of components, the current factorial experimental trial will randomize 16 geographical areas to 8 experimental conditions (cluster randomization) in each country. There will be a total of 16 groups (with 2 groups per experimental condition).

It is important to note that although there are 8 experimental conditions, this experiment should not be considered an 8-arm RCT. The purpose of this factorial experiment is to estimate the main effects of the three intervention components and interactions between the components, not to compare the 8 experimental conditions to each other. Each main effect and interaction estimate is based on all of the experimental conditions. Instead of recruiting the originally planned 240 participants per country, we will over-recruit (n = 288 per country) to account for study attrition identified in Phase 1 (https://clinicaltrials.gov/ct2/show/NCT03552250?term=Prevention+of+Child+Mental+Health+Problems+in+Southeastern+Europe+%28RISE%29&rank=1) (approx. 20-30%) in order to avoid empty cells and being at risk of being underpowered.

This study will examine the following hypotheses related to the selected components based on a conceptual model* tested in the factorial experiment:

1. Component 1: Engagement Booster. We hypothesize that providing enhanced engagement boosters (i.e., high participation incentives and communication boosters) compared to a low level of engagement boosters (i.e., low participation incentives and no communication boosters) will result in higher retention and participation of parents, which in turn will indirectly result in improvements in parenting outcomes, child behavior and other secondary outcomes (via indirect effects).
2. Component 2: Program Length. We hypothesize that those receiving the shorter length program will have higher retention and participation rates than those receiving the longer program. However, the 10-session program condition compared to the 5-session program condition will have higher dosage and therefore, we expect no difference on outcomes.
3. Component 3: Fidelity Booster. We hypothesize that higher levels of fidelity boosters (i.e., training plus structured video feedback supervision) will result in higher program fidelity which will yield larger intervention effects on primary and secondary outcomes than low levels of fidelity booster (i.e., training plus supervision on-demand).
4. We hypothesize that there will be an interaction effect between Engagement Boosters and Program Length: Program Length will interact with engagement booster and lead to greater change in primary and secondary outcomes when both components are on high level. In addition, we expect a main effect of Engagement Booster of retention and participation rates, such that regardless of Program Length, high levels of Engagement Boosters will be related to higher retention and participation rates.
5. We hypothesize that there will be an interaction effect between Fidelity Booster and Engagement Booster components, such that higher levels of Fidelity Booster and Engagement Booster will result in higher retention and participation rates than either condition alone. Higher retention and participation rates will in turn be associated with greater change in primary and other secondary outcomes.
6. There will be an interaction effect between Program Length and Fidelity Booster in which program length (i.e., 10 sessions instead of 5 sessions) in combination with higher levels of Fidelity Booster (i.e., instead of on-demand) will result in larger effect on primary and secondary outcomes than either component alone.
7. Moderators: Higher baseline levels of parental mental health symptoms and problems in the family environment will be associated with greater change on primary and secondary outcomes. Other moderators of intervention effects, such as parental age, ethnicity, and gender of the child, will be examined on an exploratory basis.
8. Economic Analyses: The objective of the economic analysis for phase 2 of this project is to explore and compare the cost-effectiveness ratios for different combinations of program components and determine the most cost-effective combinations. Cost-effectiveness ratios in terms of Euros per 1-point reduction of the CBCL subscale "Aggressive Behavior" of the PLH 2-9 program and Euros per quality-adjusted life-year (QALY) gained will be calculated to assess and compare the cost-effectiveness of different combinations of program components.

In preparation for the factorial experiment in phase 2 of this study, a 5-session version of PLH 2-9 will be developed from the original program as a potentially more affordable and more accessible program. The PLH 2-9 will include the following session contents (independent of program length): one-on-one time/child-led play; praising and rewarding children; instructions, household rules, and routines; managing difficult behaviors: ignore and consequences; reflection and moving on.

* The conceptual model will be published in a manuscript version of the study protocol (preferably open access; anticipated submission date: April 2019).

ELIGIBILITY:
Inclusion Criteria (for caregivers/parents):

1. Age 18 or older;
2. Primary caregiver responsible for the care of a child between the ages of two and nine;
3. Report elevated levels of child behavior problems for the child that he/she chooses to be part of the study (based on the Child and Adolescent Disruptive Behavior Inventory, oppositional defiant disorder subscale (8 items); scores above the mean based on normative data
4. Have lived in the same household as this child at least four nights a week in the previous month and will continue to do so;
5. Agreement of being randomized to the different conditions in the study (PLH for Children program);
6. Provision of Informed consent to participate in the full study.

Exclusion Criteria (for caregivers/parents):

Exclusion criteria for adult parents or caregivers comprise:

* any adult 1) exhibiting severe mental health problems or acute mental disabilities;
* 2) that has been referred to child protection services due to child abuse.

Inclusion Criteria (for program facilitators):

1. Age 18 or older;
2. Participate in PLH facilitator training workshop;
3. Available to deliver the entire PLH 2-9 intervention
4. Provision of Informed Consent to participate in the full study

Inclusion Criteria (for program coaches)

1. Age 18 or older;
2. Previous participation in PLH facilitator training workshop;
3. Participate in PLH coach training workshop;
4. Available to deliver coaching sessions during delivery of the PLH 2-9 intervention
5. Provision of Informed Consent to participate in the full study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 835 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-05-10 (Actual); Study Completion 2020-05-10 (Actual)

PRIMARY OUTCOMES:
Change in level of aggressive behaviour in children: Child Behavior Checklist (CBCL) 11/2-5 and 6-18, parent-report, sub-scale "Aggressive behaviour" (from the Externalizing Scale) | pre; post: approx. 7 months after pre assessment (September/October 2019); follow-up: approx. 11 months after pre assessment (January/February 2020)
  The CBCL is part of the Achenbach System of Empirically Based Assessment (ASEBA) and is available for different age ranges, including the targeted range in the present study. For Phase 2, the parent-report versions for children aged 1½-5 and 6-18 are employed. It is the most widely used instrument for assessing child behavioral and emotional symptoms. In addition to the possibility to separate behavioral from emotional symptoms, the CBCL allows for assessment in multiple languages, including Romanian, Russian, and Macedonian. The externalizing subscale raw score ranges from 0 to 48 (CBCL½-5) and 0 to 70 (CBCL6-18) with higher scores indicating more problems. The aggressive behavior subscale belongs to the externalizing scale and assess aggressive behavior (e.g., "Argues a lot"; ; raw score ranges from 0 to 38 in the CBCL ½ - 5 version and 0-36 in the CBCL 6-18 version). Items are rated on a 3-point Likert scale (2 = very true or often true of the child; 0 = not true of the child).
Change in frequency of dysfunctional parenting: Parenting Scale (PS) / self-report (shortened version); total score | pre; post: approx. 7 months after pre assessment (September/October 2019); follow-up: approx. 11 months after pre assessment (January/February 2020)
  This measure is widely used in parenting interventions across the world. The scale was designed to explicitly measure dysfunctional discipline practices in parents. Three subscales may be derived (Laxness, Overreactivity, and Verbosity). For phase 2, the subscale Verbosity is excluded due to poor performance in the pilot study, consistent with numerous other studies evaluating this subscale's psychometric properties. Each item is rated on a 7-point Likert Scale in which parents are presented with a situation and then are asked to choose between two alternative responses to a situation (1 = most effective; 7 = most ineffective; i.e., situation: "When I say my child can't do something"). For computation of the subscale scores as well as the total score, the responses on the items are averaged. We will use a modified total score (only from two subscales Laxness & Overreactivity).
Change in frequency of positive parenting and effective discipline: Parenting of Young Children Scale (PARYC) / self-report (21 items); continuous total score | pre; post: approx. 7 months after pre assessment (September/October 2019); follow-up: approx. 11 months after pre assessment (January/February 2020)
  Positive parenting behavior will be assessed using parent-report of the Parenting of Young Children Scale (PARYC, 21 items). The PARYC measures the frequency of parent behavior over the previous month. Items are summed to create a total frequency scores parenting behavior as well as for the subscales: positive parenting (7 items, e.g., "how often do you play with your child"), setting limits (7 items, e.g., "how often do you stick to your rules and not change your mind") and proactive parenting (7 items, e.g., "how often do you explain what you want your child to do in clear and simple ways"). This scale has been used in PLH trials in other countries and will allow comparison of results to those studies.

SECONDARY OUTCOMES:
Change in level of internalizing problem behavior in children: Child Behavior Checklist (CBCL) 11/2-5 (31 items) and 6-18 (32 items) parent-report, Internalizing Scale; continuous sub-scale score | pre; post: approx. 7 months after pre assessment (September/October 2019); follow-up: approx. 11 months after pre assessment (January/February 2020)
  The CBCL is part of the Achenbach System of Empirically Based Assessment (ASEBA) and is available for different age ranges, including the targeted range in the present study. For the present study, the parent-report versions for children aged 1½ - 5 and 6-18 are employed. It is the most widely used instrument for assessing child behavioral and emotional symptoms. In addition to the possibility to separate behavioral from emotional symptoms, the CBCL allows for assessment in multiple languages, including Romanian (all ages), Russian (all ages), and Macedonian (6-18 version). It is a very well validated instrument that has been used across different prevention and treatment studies. The internalizing subscale raw score ranges from 0 to 62 (CBCL/1 ½ - 5 version) and 0 to 64 (CBCL/ 6 - 18 version) with higher scores indicating more emotional problems.
Change in levels of psychological distress in parents: Depression, Anxiety, and Stress Scales - short version/ self-report (21 items); continuous total score | pre; post: approx. 7 months after pre assessment (September/October 2019); follow-up: approx. 11 months after pre assessment (January/February 2020)
  Depression, Anxiety, Stress Scales (DASS) will assess parent-report of psychological distress in parents, a 21-item scale used as a screening tool to measure depression, anxiety, and stress in adults. Caregivers report on the frequency of symptoms in the previous week using a Likert scale (0 = Never, 1 = Sometimes, 2 = Often, 3 = Always; e.g., "I felt that I had nothing to look forward to"). Total DASS scores range from 0 to 63 with subscales from 0 to 21. The DASS is a widely used measure across parenting studies including those of PLH 2-9 and will allow comparison to existing results of intervention studies in non-LMICs.
Change in frequency and incidence of child maltreatment: ISPCAN-Child Abuse Screening Tool-Intervention / self-report (16 items); main focus on continuous total score, 2nd question: any effect of intervention on any of the 3 sub-scale scores? | pre; post: approx. 7 months after pre assessment (September/October 2019); follow-up: approx. 11 months after pre assessment (January/February 2020)
  Child maltreatment will be measured using parent report of the ISPCAN Child Abuse Screening Tool-Intervention scale (ICAST-I), an adaptation of a multi-national and consensus-based survey instrument measuring parent-report the incidence and prevalence of child abuse and neglect (ICAST-P). The ICAST-P was validated in 6 LMIC and 7 languages and measures four types of abuse: physical, emotional and sexual abuse, as well as neglect. The response code for the ICAST-I was adapted to a scale from 0 to more than 8 times to assess the frequency of a certain behavior in the past month. This study will assess incidence of child maltreatment by creating dichotomous variables for physical abuse, verbal abuse, and neglect, as well as an overall indication of previous child abuse. We will also assess frequency of overall abuse by summing all of the subscales as well as for each individual subscale. Regarding emotional abuse, a 5-item-version is used. Sexual abuse is not assessed in this phase.
RE-AIM Implementation: Quality | post: approx. 7 months after pre assessment (September/October 2019)
  PLH-Facilitator Assessment Tool (PLH-FAT): Seven standard behavior categories are grouped into two scales based on the core activities and process skills. Assessment of core activities includes quality of delivery during home activity review, illustrated story discussions, and practicing skills. Assessment of process skills includes modeling skills, collaborative facilitation approach, encouragement of participation, and leadership skills. Assessment by PLH coaches not blind to allocation.
RE-AIM Reach: Enrolment rate | post: approx. 7 months after pre assessment (September/October 2019)
  Number of families who attend at least one session of the program divided by the number of families recruited into the program
RE-AIM Reach: Participation rate | post: approx. 7 months after pre assessment (September/October 2019)
  Mean attendance rate for program sessions based on those families who enrolled in the program (i.e., parents who attended at least one session). Percentage of families who enrolled in the program who attended 50% and 75% or more

OTHER OUTCOMES:
Change in levels of Intimate Partner Violence (29 items); continuous total score and 4 sub-scales (level of severity) | pre; post: approx. 7 months after pre assessment (September/October 2019); follow-up: approx. 11 months after pre assessment (January/February 2020)
  Intimate partner violence will be assessed with a screening instrument, the family maltreatment measure (Heyman et al. 2013) and an adaption of the revised Conflict Tactics Scale (CTS2S). The measure assesses adult self-report of perpetration and victimization of intimate partner physical and psychological aggression. Assessments measure the frequency of negotiation, physical assault, psychological aggression, and physical injury. Answers are coded on a 5-point Likert scale of 0 to 4, with an additional response for incidences that happened but not in the past month. This measure indicates an overall indication of IPV on a level of severity (sum of items) and prevalence (dichotomous variable indicating experience of conflict or not) as well as for each subscale. Only severity is examined here. For the current study a 9-point Likert scale of 0 to 8 is used, with an additional response for incidences that happened but not in the past month.
Change in levels of parental relationship quality: Couple Satisfaction Index / self-report (4 items); continuous total score | pre; post: approx. 7 months after pre assessment (September/October 2019); follow-up: approx. 11 months after pre assessment (January/February 2020)
  This 4 item measure assesses relationship satisfaction among intimate partners. Items are summed to create a total score. CSI-4 scores can range from 0 to 21. Higher scores indicate higher levels of relationship satisfaction. CSI-4 scores falling below 13.5 suggest notable relationship dissatisfaction.
Child and Adolescent Behavior Inventory (CABI), oppositional defiant disorder subscale (9 items) | Pre (before start of intervention)
  The CABI questionnaires assesses different types of problem behaviour in childhood and adolescence. The CABI exists of 75 items measuring different areas of psychopathology, e.g., anxiety, depression, conduct disorder or attention deficit hyperactive disorder. Eight items assess oppositional defiant disorder directed towards adults and one additional item measures if any of the eight behaviors currently cause significant problems. The sum score of the first eight items can range from 0-40 and will be used as eligibility screening tool. Respondents with scores ≥10 will be included in the Optimization Study. Higher scores indicate higher levels of symptoms.
Change in quality of life: Child Health Utility 9D (CHU9D; 9 items) | pre; post: approx. 7 months after pre assessment (September/October 2019); follow-up: approx. 11 months after pre assessment (January/February 2020)
  The CHU9D measures parent-reported child health-related quality of life. The questionnaire consists of nine dimensions (worried, sad, pain, tired, annoyed, schoolwork/homework, sleep, daily routine, activities) with five levels (e.g., 1 = "don't feel worried"; 5 = "very worried"). Higher scores indicate lower levels of quality of life. The scores of the CHU9D range from 9-45.
Cost-effectiveness / cost-analyses | pre; post: approx. 7 months after pre assessment (September/October 2019); follow-up: approx. 11 months after pre assessment (January/February 2020)
  Cost-effectiveness ratios in terms of Euros per 1-point reduction of the CBCL subscale score "Aggressive Behavior" of the PLH 2-9 program and Euros per quality-adjusted life-year (QALY) gained will be calculated to assess and compare the cost-effectiveness of different combinations of program components.
RE-AIM Reach: Recruitment rate | post: approx. 7 months after pre assessment (September/October 2019)
  Number of families who were eligible for inclusion and provided consent to participate in the program divided by the number of target population who were exposed to recruitment activities
RE-AIM Implementation: Fidelity (percentage of session activities delivered per session) | post: approx. 7 months after pre assessment (September/October 2019)
  Percentage of number of session activities delivered by facilitators (by facilitator group, implementing agency, and participating country site; facilitator fidelity check-list reports)
RE-AIM Implementation: Fidelity (mean percent of activities delivered per session) | post: approx. 7 months after pre assessment (September/October 2019)
  Average number of activities delivered divided by total number of activities per session (by facilitator group, implementing agency, and participating country site; facilitator self-reports
Change in levels of parental stress: Parental Stress Scale (18-items) | pre; post: approx. 7 months after pre assessment (September/October 2019); follow-up: approx. 11 months after pre assessment (January/February 2020)
  The Parental Stress Scale measures parental stress across different domains (rewards, stressors, satisfaction, loss of control) with 18 items. An example, from the domain stressors, is "The major source of stress in my life is my child(ren)". Caregivers answer on a scale from strongly disagree (1) to strongly agree (5). The overall score ranged from 18 to 90 with higher scores indicating more parental stress.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Foran, Prof., Principal Investigator — University of Klagenfurt; Jamie Lachman, Dr., Principal Investigator — University of Oxford; Frances Gardner, Prof., Principal Investigator — University of Oxford; Judy Hutchings, Prof., Principal Investigator — Bangor University; Adriana Baban, Prof., Principal Investigator — Babes Boylai University; Marija Raleva, Prof., Principal Investigator — Institute for Marriage, Family and Systemic Practice - ALTERNATIVA; Galina Lesco, Dr., Principal Investigator — Health for Youth Association, Moldova; Catherine Ward, Prof., Principal Investigator — University of Cape Town; Xiangming Fang, Prof., Principal Investigator — Georgia State University
Locations (3):
- Health for Youth Association, Chisinau, Moldova
- Institute for Marriage, Family and Systemic Practice - ALTERNATIVA, Skopje, North Macedonia
- Babes Boylai University, Cluj-Napoca, Romania

IPD SHARING:
Plan to Share IPD: Yes
It is planned to share results to members of the scientific community with an interest in parenting interventions, behavioral problems in children, process evaluation, the transferability of interventions across cultures and contexts, and the MOST (the Multiphase Optimization Strategy). The aim is to sustain the intervention after the end of the project by including local authorities, policy makers, and other stakeholders such as community groups and caregivers in the intervention from each country. Further, we will archive the dataset and upload metadata in the certified repository Zenodo at https://zenodo.org/. Further details about IPDSharing are described in the Data Management Plan and this is available by contacting Prof. Heather Foran (heather.foran@aau.at).
Supporting Information: Study Protocol
Time Frame: Study Protocol will be shared once it is published (preferably open access)
Access Criteria: (see above)

REFERENCES:
- [Background] Barlow J, Johnston I, Kendrick D, Polnay L, Stewart-Brown S. Individual and group-based parenting programmes for the treatment of physical child abuse and neglect. Cochrane Database Syst Rev. 2006 Jul 19;(3):CD005463. doi: 10.1002/14651858.CD005463.pub2. PMID 16856097
- [Background] Chen M, Chan KL. Effects of Parenting Programs on Child Maltreatment Prevention: A Meta-Analysis. Trauma Violence Abuse. 2016 Jan;17(1):88-104. doi: 10.1177/1524838014566718. Epub 2015 Jan 8. PMID 25573846
- [Background] Knerr W, Gardner F, Cluver L. Improving positive parenting skills and reducing harsh and abusive parenting in low- and middle-income countries: a systematic review. Prev Sci. 2013 Aug;14(4):352-63. doi: 10.1007/s11121-012-0314-1. PMID 23315023
- [Background] Mikton, C. (2012). Two challenges to importing evidence-based child maltreatment prevention programs developed in high-income countries to low- and middle-income countries: Generalizability and affordability. In H. Dubowitz (Ed.), World perspectives on child abuse (p. 97). Aurora, CO: International Society for the Prevention of Child Abuse and Neglect.
- [Derived] Bruhl A, Waller F, Foran HM, Jansen E, Hutchings J, Heinrichs N. Spillover mechanisms linking intimate partner violence and child maltreatment: a cross-sectional and longitudinal study among Eastern European mothers. BMC Public Health. 2025 Nov 4;25(1):3778. doi: 10.1186/s12889-025-24955-8. PMID 41188856
- [Derived] Frantz I, Foran HM, Lachman JM, Gardner F, McMahon RJ, Ogden T, Hutchings J, Costin MR, Kunovski I, Raleva M, Mueller J, Heinrichs N. Adverse event assessment in a parenting programme: experiences from a multisite randomised controlled trial. Trials. 2024 Aug 17;25(1):547. doi: 10.1186/s13063-024-08357-6. PMID 39154169
- [Derived] Lachman JM, Heinrichs N, Jansen E, Bruhl A, Taut D, Fang X, Gardner F, Hutchings J, Ward CL, Williams ME, Raleva M, Baban A, Lesco G, Foran HM. Preventing child mental health problems through parenting interventions in Southeastern Europe (RISE): Protocol for a multi-country cluster randomized factorial study. Contemp Clin Trials. 2019 Nov;86:105855. doi: 10.1016/j.cct.2019.105855. Epub 2019 Oct 24. PMID 31669446
- See also: Project website — http://www.rise-plh.eu/index.html